CLINICAL TRIAL: NCT03363282
Title: Recurrence Rate of Mini-SLET (Simple Limbal Epithelial Transplantation) vs. Limbal-Conjunctival Autograft in Primary Pterygium Excision
Brief Title: Recurrence Rate of Mini-SLET vs. Limbal-Conjunctival Autograft in Primary Pterygium Excision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CI-021-2015
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Pterygium of Conjunctiva and Cornea
Keywords: Crosslinking
MeSH Terms: conditions — Pterygium Of Conjunctiva And Cornea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mini-SLET (Experimental): Simple Limbal Epithelial Transplantation
  Interventions: Procedure: Pterygium Excision
- Limbal-Conjunctival Autograft (Experimental): Patients treated with limbal-conjunctival autograft
  Interventions: Procedure: Pterygium Excision

INTERVENTIONS:
Procedure: Pterygium Excision — Pterygium excision is the first step for repair
  Other Names: Limbal-Conjunctival Autograft; Mini-SLET

SUMMARY:
To study the efficacy and safety of amniotic membrane transplantation as an adjunctive therapy after surgical excision of primary pterygium and compare the clinical outcomes with conjunctival autograft

DETAILED DESCRIPTION:
Prospective Randomized Blind Clinical Trial

Sixty-four eyes of 64 patients with primary nasal pterygium have been operated by two surgeons (E. G-H, A. N-C). All patients are randomized to undergo Mini-SLET or limbal-conjunctival autograft transplantation as an adjuvant therapy after pterygium excision.

Four eyes were treated with Mini-SLET(group 1), and 26 eyes have been operated with conjunctival autograft (group 2). Patients will be followed up at 1 day, 1 week, 1, 3, 6, 9 and 12 months postoperation. The main outcome measurement was a recurrence rate after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary nasal pterygium > 2mm

Exclusion Criteria:

* Pregnant
* Previous ocular surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2016-11-17 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Recurrence rate | one day
  Regrowth of pterygium

IPD SHARING:
Plan to Share IPD: No
Patient data will be analyzed by a single researcher

REFERENCES:
- [Result] Tseng SC. Concept and application of limbal stem cells. Eye (Lond). 1989;3 ( Pt 2):141-57. doi: 10.1038/eye.1989.22. PMID 2695347
- [Result] Tananuvat N, Martin T. The results of amniotic membrane transplantation for primary pterygium compared with conjunctival autograft. Cornea. 2004 Jul;23(5):458-63. doi: 10.1097/01.ico.0000116522.57227.97. PMID 15220729
- [Result] Kucukerdonmez C, Akova YA, Altinors DD. Comparison of conjunctival autograft with amniotic membrane transplantation for pterygium surgery: surgical and cosmetic outcome. Cornea. 2007 May;26(4):407-13. doi: 10.1097/ICO.0b013e318033b3d4. PMID 17457187
- [Derived] Oliva-Bienzobas V, Nava-Castaneda A, Jimenez-Corona A, Kahuam-Lopez N, Ramirez-Miranda A, Navas A, Graue-Hernandez EO. Comparison of mini-simple limbal epithelial transplantation and conjunctival-limbal autograft for the treatment of primary pterygium: a randomised controlled trial. Br J Ophthalmol. 2023 Nov 22;107(12):1776-1781. doi: 10.1136/bjo-2021-320707. PMID 37739769